CLINICAL TRIAL: NCT04443491
Title: Estimating the Transpulmonary Pressure From the Central Venous Pressure in Mechanically Ventilated Patients With Respiratory Failure
Brief Title: Comparison of Esophageal and Central Venous Pressure for Estimating Transpulmonary Pressure Changes
Acronym: PPLproject
Status: Completed | Type: Observational
Sponsor: University of Siena (Other)
Responsible Party: Principal Investigator, Federico Franchi, Principal Investigator; Associate professor of Anesthesiology; Anesthesia and Intensive Care Unit, Department of Medicine, Surgery and Neuroscience, University of Siena, Siena, Italy, University of Siena
Other Study IDs: PPL project
Record Dates: First submitted 2020-06-01; First posted 2020-06-23 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Mechanical Ventilation; Acute Respiratory Distress Syndrome
Keywords: esophageal pressure; transpulmonary pressure; central venous pressure; acute respiratory failure
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Central venous pressure (CVP) is characterized by a low-frequency pleural-dependent as well as a high-frequency cardiac pulsatile component. The aim of the study is to compare the low-frequency component of CVP with the esophageal pressure (Pes), as surrogate of pleural pressure, to estimate trans-pulmonary pressure (PL).

DETAILED DESCRIPTION:
The investigators will enroll mechanically ventilated patients admitted to the intensive care unit with the diagnosis of respiratory failure monitored with a dedicated nasogastric catheter and a central venous catheter for measuring Pes and CVP, respectively. Electrocardiogram trace, Pes, CVP and airway pressure (Paw) will be recorded at the end of inspiratory and expiratory pauses. The CVP waveforms will be analyzed off-line using a dedicated low-pass digital filter to obtain the low-frequency component of CVP (filtered CVP, fCVP). Paw, Pes and fCVP will be used to calculate PL using transpulmonary driving pressure formula (PL-Pes and PL-fCVP, respectively). The PL values obtained with fCVP and Pes will be compared to assess the correlation of the two methods.

ELIGIBILITY:
Inclusion Criteria:

* adult patients receiving invasive mechanical ventilation
* diagnosis of acute respiratory failure (defined as the ratio of partial oxygen pressure and fraction of inspired oxygen below 200 mmHg)
* esophageal balloon catheter
* central venous catheter

Exclusion Criteria:

* age under 18 years old
* Hemodynamic instability
* Esophageal diseases (varices, stenosis..)
* Refusal of the patient
* evidence of active air leak from the lung (pneumothorax, pneumomediastinum, existing chest tube....)
* history of lung/abdominal surgery
* pregnancy
* severe coagulopathy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to ICU treated with mechanical ventilation.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Transpulmonary pressure | Within 72 hours from the starting of mechanical ventilation
  Correlation and agreement between the transpulmonary pressure obtained from esophageal balloon catheter and central venous catheter

SECONDARY OUTCOMES:
Transpulmonary pressure in subgroups of patients | Within 72 hours from the starting of mechanical ventilation
  Agreement between trans pulmonary pressure obtained with the two methods in subgroup of patients such as those with acute respiratory distress syndrome or obesity
Transpulmonary pressure in patients at risk for ventilator-induced-lung-injury | Within 72 hours from the starting of mechanical ventilation
  Comparison of the transpulmonary pressure obtained with the two methods in patients at risk for ventilator-induced-lung-injury

CONTACTS AND LOCATIONS:
Overall Officials: Federico Franchi, MD, Principal Investigator — University of Siena, Depatment of Medical Biotechnology
Locations (1):
- Azienda Ospedaliera Universitaria Senese, Siena, Italy

IPD SHARING:
Plan to Share IPD: No